CLINICAL TRIAL: NCT05303909
Title: The Immunostimulatory Effects of Gentamicin: Translating Aminoglycoside Antibiotics Into Antiviral Therapeutics for Pandemic Response (Part B)
Brief Title: The Immunostimulatory Effects of Gentamicin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment due to COVID19
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GENT-YF-01B
Record Dates: First submitted 2022-03-13; First posted 2022-03-31 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
Keywords: Gentamicin; viremia; YF17D
MeSH Terms: conditions — Viremia | interventions — Gentamicins

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to receive either a single dose of IV gentamicin at dose of 5 mg/kg or 0.9% normal saline placebo on Day 0 in a double-blind fashion, followed by YF17D vaccination 30 minutes later.
Who Masked: Participant, Investigator
Masking Description: This is a double blind placebo controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentamicin (Experimental): a single dose of IV gentamicin at a dose of 5 mg/kg (rounded up to the nearest 10mg) diluted in 100mls of 0.9% normal saline infused over 30 minutes via a peripheral vein
  Interventions: Drug: Gentamicin
- Placebo (Placebo Comparator): 100mls of 0.9% normal saline as placebo infused over 30 minutes via a peripheral vein
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gentamicin — a single dose of IV gentamicin at a dose of 5 mg/kg infused over 30 minutes via a peripheral vein. Followed by administration of YF17D vaccine (stamaril) 0.5mls via subcutaneous injection into the deltoid region of the right or left arm.
  Arms: Gentamicin
Drug: Placebo — 100mls of 0.9% normal saline as placebo infused over 30 minutes via a peripheral vein. Followed by administration of YF17D vaccine (stamaril) 0.5mls via subcutaneous injection into the deltoid region of the right or left arm.
  Arms: Placebo

SUMMARY:
Gentamicin is one of the few aminoglycoside antibiotics which are approved for parenteral use in Singapore. As with other aminoglycosides, gentamicin is primarily bactericidal against Gram-negative organisms. It is well known that viral infection increases susceptibility to bacterial infection; increased rates of Gram-negative bacterial sepsis due to gastrointestinal tract bacterial translocation have been reported in Ebola and dengue patients. Gentamicin use in viral infection could thus improve clinical outcome by inhibiting both viral and opportunistic Gram-negative bacterial infection.

Parenteral aminoglycosides do not cause perturbations or dysbiosis within the human gut microbiome. This is of importance as dysbiosis would not only increase the risk of antibiotic-resistant bacteria selection within the intestinal tract, it could also lead to negative downstream effects on the host response to infection by altering activation states of both innate and adaptive immunity. Thus, parenteral gentamicin may offer a unique approach to preventing both viral and downstream secondary Gram-negative bacterial infection, while at the same time minimizing the potential development of antibiotic resistance.

The overarching goal of this study is to demonstrate that parenteral aminoglycosides exert broad-spectrum antiviral effects against RNA viruses in humans through their immunostimulatory properties. Using the live attenuated yellow fever (YF17D; stamaril) vaccine as an experimental viral infection model, a placebo controlled clinical trial will be carried out to demonstrate the efficacy of parenteral gentamicin in preventing viremia.

DETAILED DESCRIPTION:
Informed written consent will be sought from subjects who fulfil criteria for enrolment. All consented subjects will undergo screening, which includes physical examination, full blood count, liver function test, serum creatinine, and urinary pregnancy test (for female subjects of child-bearing potential).

All eligible subjects will proceed to Day 0, where they will undergo randomization to receive either IV gentamicin at a dose of 5 mg/kg or 0.9% normal saline placebo, followed by YF17D vaccination 30 minutes later i.e. 30 minutes after completion of gentamicin/placebo infusion. Urine pregnancy test (for female subjects of child-bearing potential) will be performed prior to study drug administration. Baseline physical examination and vital signs will be done as well. On Day 0, research blood sampling will be performed prior to gentamicin/placebo administration.

Subsequently, study subjects will return for follow-up visits on D1, D4, D6, D14 and D30. Research blood samples will be taken at each visit. Physical examination, vital signs, and review of adverse events will be done at each of the visit as well.

At any time post-study drug or YF17D administration, subjects will be trained to observe for systemic AEs. A diary will also be given to the subjects to record such events should they occur during this period. Should they develop systemic symptoms that require intervention, they will report to the study site for medical evaluation and receive the appropriate therapy. Duration of symptoms will be recorded. Any concomitant medication use during this period will also be recorded.

During the study, full history taking and physical examination will be performed at both scheduled and unscheduled visits. The Common Terminology Criteria for Adverse Events (CTCAE), routinely employed in clinical trials, will be used to define AE terminology and severity. Management of AEs is at the discretion of the study team PI and co-Is, guided by severity and clinical indication for intervention. All medication prescribed for the management of AEs will be documented in the medication/concomitant medication clinical record form.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, 21-50 years of age at time of screening
2. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. The laboratory values must be within the normal range of the assessing site or show abnormalities that are deemed not clinically significant as judged by the investigator. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event.
3. Accessible vein for blood collection.
4. Subjects who are willing to comply with the requirements of the study protocol and scheduled visits. (e.g. return for follow-up visits) and who are willing to make themselves available for the duration of the study, with access to a consistent means of telephone contact, which may be either at home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device (i.e. a common-use phone serving multiple rooms or apartments).
5. Ability to provide informed consent
6. Female subjects of non-child bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Post-menopausal subjects must have had at least 12 months of natural (spontaneous) amenorrhea.
7. Female subjects of childbearing potential with negative urine pregnancy tests on the day of screening and day of antibiotic administration.
8. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) must agree to use adequate and reliable contraceptive measures (e.g. spermicides, condoms, contraceptive pills) or practice abstinence for 10 days after vaccination

Exclusion Criteria:

1. History of presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, haematological, endocrine or immunosuppressive disorders that would be a risk factor when administered gentamicin or YF17D vaccine.
2. Previous receipt of YF17D vaccine (stamaril) or any other yellow fever vaccines.
3. Previous history of Yellow fever virus infection
4. Known allergy to YF17D vaccine (stamaril) or its components
5. Known allergy to gentamicin
6. History of severe food/drug/vaccine allergies e.g. angioedema, anaphylaxis
7. Known allergy to egg or egg products
8. History of thymus gland disease
9. Diagnosed with cancer or on treatment for cancer (with the exception of localized basal cell carcinoma) within 3 years prior to screening
10. Diagnosed with neuromuscular disorders
11. Evidence of clinically significant anemia (Hb <10 g/dl)
12. Blood donation exceeding >450mls in the past 3 months
13. Presence of acute infection in the preceding 7 days or presence of a temperature ≥ 38.0°C (oral or tympanic temperature assessment), or acute symptoms greater than of "mild" severity on the scheduled date of first dose
14. Woman who is pregnant or breast feeding
15. Evidence of substance abuse, or previous substance abuse including alcohol
16. Participation in a study involving administration of an investigational compound (including investigational vaccines) within the past three months, or planned participation during the duration of this study.
17. Receipt of anti-inflammatory drugs (such as NSAIDs or steroids) in the past 7 days before the first study drug/vaccine dose.
18. Receipt of any licensed vaccine in the past 30 days before the first study drug/vaccine dose.
19. Any condition that, in the opinion of the investigator, would complicate or compromise the study or wellbeing of the subject.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with detectable YF17D viremia | 14 days
  The proportion of subjects with detectable YF17D viremia after YF17D vaccination

SECONDARY OUTCOMES:
Peak YF17D viremia levels | 14 days
  Peak YF17D viremia levels after YF17D vaccination
Duration of detectable YF17D viremia | 14 days
  Duration (in days) of detectable YF17D viremia after YF17D vaccination
Neutralising antibody titers against YF17D | 30 days
  Neutralising antibody titers at study Day 30 against YF17D after YF17D vaccination
Rates of symptomatic infection after YF17D vaccination | 30 days
  Rates of symptomatic infection after YF17D vaccination
Levels of innate immune gene expression | 6 days
  Levels of innate immune gene expression in subjects.
Mean YF17D viremia levels | 14 days
  Mean YF17D viremia levels after YF17D vaccination

OTHER OUTCOMES:
Cellular immune response | Day 30
  Levels of Cellular immune response (Spot Forming Units as measured by T cell EliSPOT) in subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided